CLINICAL TRIAL: NCT06848231
Title: A Double-Blind, Placebo-Controlled, Multi-Center, Phase II, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of YA-101 in Subjects With Multiple System Atrophy
Brief Title: A Phase 2 Study of YA-101 in Patients With Multiple System Atrophy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yoda Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YA-101-201
Record Dates: First submitted 2025-02-17; First posted 2025-02-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-06

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- YA-101 (Experimental)
  Interventions: Drug: YA-101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YA-101 — Drug: YA-101
  • YA-101 taken BID
  Arms: YA-101
Drug: Placebo — Placebo taken BID
  Arms: Placebo

SUMMARY:
This is a Phase 2, double-blind, placebo-controlled, multi-center, Phase II, dose escalation study to evaluate the safety, tolerability, pharmacokinetics and efficacy of Ya-101 in subjects with multiple system atrophy.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate 2 doses of YA-101 compared to placebo in MSA patients, including: 1) safety and tolerability, 2) pharmacokinetics, and 3) potential efficacy of YA-101.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the process of the clinical trial and give informed consent for the participation of the study.
2. Diagnosis of MSA according to MDS clinical criteria (Wenning et al, 2022), including subjects with MSA of either subtype (MSA-P or MSA-C).
3. Males or non-pregnant, non-lactating females with no child-bearing potential, or agree to use 2 forms of contraception.
4. Able to take oral medications.
5. Able to ambulate without the assistance of another person.

Exclusion Criteria:

1. Positive urine test for drugs of abuse and/or alcohol test both at screening and Day 1.
2. Evidence of renal impairment or hepatic impairment.
3. Subject with a Mini-Mental State Examination (MMSE) score of 24 or lower.
4. Medical history includes severe systemic diseases such as cardiopulmonary failure, severe liver or kidney disease, and uncontrolled diabetes; significant central nervous system disorders like stroke, encephalitis, and epilepsy and severe head trauma; peptic ulcer in one year prior to screening.
5. Positive results for active viral infections, including human immunodeficiency virus (HIV), hepatitis B, and hepatitis C.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | Baseline to Day 112
  Incidence and severity of Adverse Events (AEs).

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | Baseline to Day 84
  To describe the pharmacokinetics parameter (Cmax) of YA-101 using sparse PK sampling.
Area under the concentration-time curve (AUC) | Baseline to Day 84
  To describe the pharmacokinetics parameter (AUC) of YA-101 using sparse PK sampling.
Time of maximum observed concentration (Tmax) | Baseline to Day 84
  To describe the pharmacokinetics parameter (Tmax) of YA-101 using sparse PK sampling.
Change from baseline in Unified Multiple System Atrophy Rating Scale (UMSARS) over time | Baseline to Day 112
  The unified multiple system atrophy rating scale (UMSARS) is composed of four subscales: UMSARS-I (12 items) rates patient-reported functional disability, UMSARS-II (14 items) assesses motor impairment based on a clinical examination, UMSARS-III records blood pressure and heart rate in the supine and standing positions, and UMSARS-IV (1 item) rates chore-based disability. Higher scores on the UMSARS indicate greater disability.
Change from baseline in the 10-meter walking test | Baseline to Day 112

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - UCLA Health, Los Angeles, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University Irving medical center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Juntendo University Hospital, Tokyo, Japan
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: Undecided